CLINICAL TRIAL: NCT02180685
Title: Reconstruction of the Medial Patellofemoral Ligament - A Randomised Controlled Trial Comparing Two Surgery Technics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Danish EC 1-10-72-194-14
Record Dates: First submitted 2014-06-30; First posted 2014-07-03 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Knee Stability; Patella Luxation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anchor fixation (Other): Medial fixation of the reconstruction at the medial femural condyle with suture anchors.
  Interventions: Other: Anchor fixation
- Screw fixation (Other): Medial fixation of the reconstruction at the medial femural condyle with a screw.
  Interventions: Other: Anchor fixation

INTERVENTIONS:
Other: Anchor fixation

SUMMARY:
The purpose of this present study is to determine which surgery technic provides the best clinical outcome after medial patellofemoral ligament reconstruction comparing suture anchors and screw fixation in medial femoral condyle.

ELIGIBILITY:
Inclusion Criteria:

* patella luxation, more than 2 times

Exclusion Criteria:

* cartilage damage (grad 3)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of subjective symptoms with a patient reported outcome score | Baseline, 6 months 12 Months, 24 months
  Anterior Knee Pain Scale

SECONDARY OUTCOMES:
Patient reported outcome scores | Baseline, 6 months 12 Months, 24 months
  Tegner
Patient reported outcome scores | Baseline, 6 months 12 Months, 24 months
  KOOS (Knee injury and osteoarthritis outcome score)
Re-operation rate | Baseline, 6 months 12 Months, 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Trauma, Tage-Hansens Gade 2b, Aarhus, Denmark